CLINICAL TRIAL: NCT02883140
Title: Prospective, Pilot, Comparative, Monocentric Study of Diagnosis Capabilities of the Three-dimensional Cone-Beam CT Sialography (3D-CBCT Sialography) and MRI Sialography in Non-tumor Salivary Diseases
Brief Title: Imaging Study of 3D-CBCT Sialography and MRI Sialography in Non Tumor Salivary Diseases
Acronym: PIGS
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC15_0196
Record Dates: First submitted 2016-05-10; First posted 2016-08-30 (Estimated); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Non Tumor Salivary Gland Diseases of the Parotid Glands; Non Tumor Salivary Gland Diseases of the Submandibular Glands
Keywords: Sialography; Cone-beam CT; MRI sialography; non tumor salivary symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Three-dimensional sialography CBCT and MRI sialography — 1. MRI sialography: Achieved on a 3 Tesla MRI (INGENA 3T Philips Medical Systems). Patient supine positioned. Sialo-MR sequences (3D T2 DRIVE, TSE, SENSE and SPIR) and conventional sequences (T2 turbo spin echo).
  2. 3D CBCT sialography: Achieved same day as the MRI sialography, after acute episode subsided. 0.5ml of high concentration, water-soluble, iodinated contrast product (HEXABRIX 320®, 320g /L, Guerbet, France) is injected in the symptomatic salivary gland and maintained in the gland. Image acquisition performed on a wide-field CBCT device (NewTom VGi, QR, Verona, Italy). Front and profile scout views achieved. mA and exposure time modulated according to scout views. Reconstruction in Maximal Intensity Projection, 3-dimensional and MultiPlanar Reconstructions sections

SUMMARY:
Non tumor salivary gland diseases are common and include sialadenitis, sialadenosis, stones, stricture and ductal dilatation, anatomical abnormalities. A radiological examination is required in order to sign the diagnosis, locate precisely the lesions and define the therapeutic strategy. Cone beam computerized tomography (CBCT), because of its accessibility and the possibilities it offers in terms of image processing, is a potential alternative to the conventional sialography and to the MRI sialography, considered as a gold standard procedure. Our comparative study, aims to evaluate the diagnostic performance of the 3D-CBCT sialography compared to MRI sialography, in patients with non tumor ductal salivary diseases.

DETAILED DESCRIPTION:
Our study focuses on patients over 18 years, with unilateral or bilateral parotid or submandibular salivary symptoms. Each patient included is given a MRI sialography and a 3D-CBCT sialography at a later stage when the acute episode has subsided. Images are archived on the Carestream Picture Archiving Communication System (PACS). Interpretation is achieved after Multi-Planar Reconstruction (MPR), Maximal Intensity Projection (MIP) and three-dimensional rendering. A primary radiological analysis of the two procedures is systematically done by a specialist radiologist for the diagnostic and therapeutic care of the patient. A second radiological data analysis is carried out at the end of the study, by a specialized radiologist, different from the first one, to asses the two radiological examinations.

The primary outcome measure is the capability of the radiological technique to detect a ductal salivary feature. Secondary outcomes include the clinical characteristics of the patients, the diagnostic capabilities in identifying the salivary lesions, their number, their precise location and measurements. A primary side effect in catheterization and dosimetric parameters for the CBCT technique will be systematically recorded.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, over 18 years old.
* With unilateral or bilateral parotid or submandibular salivary symptoms (salivary swelling, salivary colic, pain, salivary infections), with an acute evolution (<14 days), subacute (2-12 weeks) or chronic one (>3 months).
* With or without initial imaging (ultrasonography).
* Understanding the technique and its interest in the diagnostic and therapeutic management.
* Accepting the examination and the salivary catheterization.
* Positive catheterization test

Exclusion Criteria:

* Patient whose physical or mental condition make him unable to understand the examination and to consent to the study.
* Allergy to iodine.
* Salivary infection under treatment.
* Damage to the oral mucosa preventing salivary catheterization.
* Contraindication to MRI: metal or valvular prosthesis, pacemaker, claustrophobia.
* Current or suspected pregnancy.
* Patient refusing the examination or the catheterization.
* Salivary symptoms of tumor appearance: Unilateral palpable mass, facial palsy, multiple lymph nodes in parotid and / or pre-auricular and / or neck areas.
* Salivary neoplasm demonstrated by a prior diagnostic testing.
* Patient who underwent head and neck scan in the previous 6 months. Conventional or three dimensional sialography achieved in the previous 6 months.
* Salivary catheterization failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female, over 18 years old with unilateral or bilateral parotid or submandibular salivary symptoms (salivary swelling, salivary colic, pain, salivary infections), with an acute evolution (<14 days), subacute (2-12 weeks) or chronic one (>3 months)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2019-08-18 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Detection of a salivary ductal disease with the 3D-CBCT sialography and the MRI sialography: Yes/No. | 1 day

SECONDARY OUTCOMES:
Precise location of lesions in the ductal system, identified as CSx for the Stensen's duct divisions and CWx for the Wharton's duct divisions (where CS1 and CW1 correspond to the main Stensen's and Wharton's ducts respectively) | 1 day
Identification of the last salivary duct division visualized, identified as CSx for the Stensen's duct divisions and CWx for the Wharton's duct divisions | 1 day
Operational safety: Looking for adverse effects of the catheterization (pain, bleeding, ductal perforation) | 1 day
Dose Area Product (mGy.cm-2) for 3D-CBCT sialography | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Delemazure Anne-Sophie, MD, Principal Investigator — Nantes University Hospital

IPD SHARING:
Plan to Share IPD: Undecided
Not applicable now.

REFERENCES:
- [Derived] Bertin H, Bonnet R, Le Thuaut A, Huon JF, Corre P, Frampas E, Langlois EM, Chesneau AD. A comparative study of three-dimensional cone-beam CT sialography and MR sialography for the detection of non-tumorous salivary pathologies. BMC Oral Health. 2023 Jul 8;23(1):463. doi: 10.1186/s12903-023-03159-9. PMID 37420227